CLINICAL TRIAL: NCT03193255
Title: Efficacy and Safety of Povidone Iodine-based Disinfecting Solution (cleadewGP) for Rigid Contact Lenses
Brief Title: Efficacy and Safety of cleadewGP for Rigid Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Ophtecs Corporation (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20170430002
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Contact Lens Solution Toxicity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No daily lens rubbing (Active Comparator): Daily lens disinfection with OPHTECS cleadew GP without lens rubbing
  Interventions: Device: OPHTECS cleadew GP
- Daily rubbing (Active Comparator): Daily lens disinfection with OPHTECS cleadew GP after lens rubbing with cleadew GP
  Interventions: Device: OPHTECS cleadew GP
- Daily rubbing with separate cleaner (Active Comparator): Daily lens disinfection with OPHTECS cleadew GP after lens rubbing with a daily lipid cleaner
  Interventions: Device: OPHTECS cleadew GP
- Daily rubbing and weekly protein removal (Active Comparator): Daily lens disinfection with OPHTECS cleadew GP after daily lipid cleaner followed by weekly protein removal treatment
  Interventions: Device: OPHTECS cleadew GP

INTERVENTIONS:
Device: OPHTECS cleadew GP — Povidone-iodine based disinfecting solutions for rigid contact lenses

SUMMARY:
Multipurpose solutions (MPS) are the most commonly prescribed regimen to clean, disinfect and rinse rigid lenses. The preservatives used in MPS may cause hypersensitivity and the presence of quaternary ammonium compounds (QAC) may increase development of antiseptic resistance mediated by QAC resistance genes, thus lowering the efficacy of disinfection. Povidone-iodine (PVI) has been safely used as a disinfectant for ophthalmic operations and eye drops. The cleadew GP (Ophtecs, Japan) tested in the current study is a PVI based rigid lens disinfecting solutions which does not employ QAC. If its efficacy and safety can be confirmed in this study, it will be a good alternative rigid lens care regimen for children.

DETAILED DESCRIPTION:
Multipurpose solutions (MPS) are the most commonly prescribed regimen to clean, disinfect and rinse rigid lenses. These solutions usually contain quaternary ammonium compounds (QAC) which have been shown to be selective for carriage of organisms harbouring QAC genes in orthokeratology (ortho-k) lens wear and it raises concerns about safety with the increasing popularity of orthokeratology (ortho-k) for myopia control in children. Hydrogen peroxide system is a good alternative but this option is limited in rigid lens market. The only brand available in Hong Kong labelled as safe for rigid contact lenses has limited disinfecting power. cleadewGP (Ophtecs, Japan) is a new disinfecting solution for rigid contact lenses which does not employ QAC and instead is povidone iodine (PVI) based. PVI has been safely used as a disinfectant for ophthalmic operations and is commonly used in eye drops. PVI-based soft and rigid lens solutions have been reported to be as effective against Pseudomonas aeruginosa as other MPS and hydrogen peroxide-based solutions. However, other efficacy against other organisms need to be demonstrated to allow this solution to meet FDA requirements. The PVI-based soft lens solution was also reported to be effective against Acanthamoeba. cleadewGP is relatively new in the market and not much work has been done on the efficacy and safety of this solution. If confirmed to be effective and safe, cleadewGP may be a better alternative to ortho-k lens wearers who need to use disinfecting solutions at least for a few years while under ortho-k treatment. In the absence of QAC, there will be no concern of selection of carriage of organisms harbouring QAC genes in ortho-k lens wearers using this disinfecting solution over time.

The current study aims at investigating the effectiveness and safety of the cleadewGP for cleaning (lipid and protein removal) and disinfecting of ortho-k lenses by comparing the outcomes collected from subjects randomly assigned to one of the following study groups.

Group 1: cleadewGP without lens rubbing Group 2: cleadewGP with lens rubbing Group 3: cleadewGP with separate daily cleaner Group 4: cleadewGP with separate daily cleaner and weekly protein removal agent

Four study visits will be involved in this 6 months study: baseline, 1-month, 3-month, and 6-month after lens wear. Complimentary solutions will be provided during the study period. Solutions and accessories will be replaced at monthly interval. Effectiveness for cleaning and disinfection and safety of lens wear will be determined by comparing the changes in ocular microbiome before and after lens wear, contamination levels of lenses and accessories, biomicroscopic examination of lenses and eyes, and subjective rating of lens comfort among the four groups of subjects.

ELIGIBILITY:
Inclusion Criteria:

* cycloplegic objective sphere between -1.00D to -4.00D
* cycloplegic objective astigmatism ≤ 2.00D
* anisometropia < 1.00D
* best-corrected logMAR visual acuity 0.10 or better in both eyes
* symmetrical corneal topography with toricity ≤ 2.00D
* normal ocular health

Exclusion Criteria:

* contraindication to ortho-k wear
* prior history of myopia control treatment
* prior history of rigid contact lens wear
* strabismus or amblyopia
* systemic or ocular conditions which might affect refractive development
* poor response or poor compliance to lens wear including poor lens handling, poor vision, and/ocular response after lens modifications

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in subjective symptoms before and 6 months after lens wear | 6 months
  Questionnaire of ocular comfort will be administered to rate symptoms of discomfort, itching, tearing, dryness and redness
Change in corneal staining and injection before and 6 months after ortho-k lens wear | 6 months
  Grading of corneal staining, limbal injection and conjunctival injection under slitlamp biomicroscopy before and after ortho-k lens wear

SECONDARY OUTCOMES:
Change in levels of ocular microbiome before and 6 months after ortho-k lens wear | 6 months
  Sample from the lower conjunctiva will be gently taken with cotton swab pre-wet with normal saline before and ortho-k lens wear
Levels of contamination of lens cases | 6 months
  Sample will be collected from the left compartment of the lens case to determine the presence of microorganisms. The right compartment of the lens case will be tested for the presence and amount of biofilm
Levels of contamination of lenses | 6 months
  Samples will be collected from the left lens surface to test for the presence of microorganisms

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi GS, Boost M, Cho P. Prevalence of antiseptic-resistance genes in staphylococci isolated from orthokeratology lens and spectacle wearers in Hong Kong. Invest Ophthalmol Vis Sci. 2015 May;56(5):3069-74. doi: 10.1167/iovs.15-16550. PMID 25788652
- [Background] Guang-Sen S, Boost M, Cho P. Prevalence of antiseptic resistance genes increases in staphylococcal isolates from orthokeratology lens wearers over initial six-month period of use. Eur J Clin Microbiol Infect Dis. 2016 Jun;35(6):955-62. doi: 10.1007/s10096-016-2622-z. Epub 2016 Mar 18. PMID 26993290
- [Background] Trinavarat A, Atchaneeyasakul LO. Treatment of epidemic keratoconjunctivitis with 2% povidone-iodine: a pilot study. J Ocul Pharmacol Ther. 2012 Feb;28(1):53-8. doi: 10.1089/jop.2011.0082. Epub 2011 Sep 14. PMID 21916618
- [Background] Isenberg SJ. The ocular application of povidone-iodine. Community Eye Health. 2003;16(46):30-1. No abstract available. PMID 17491857
- [Background] Rampat R, Jain S. The effect of commonly used surgical solutions on the tensile strength of sutures. J Pediatr Ophthalmol Strabismus. 2014 May-Jun;51(3):189-90. doi: 10.3928/01913913-20140318-01. Epub 2014 Mar 25. PMID 24654799
- [Background] Martin-Navarro CM, Lorenzo-Morales J, Lopez-Arencibia A, Valladares B, Pinero JE. Acanthamoeba spp.: efficacy of Bioclen FR One Step, a povidone-iodine based system for the disinfection of contact lenses. Exp Parasitol. 2010 Sep;126(1):109-12. doi: 10.1016/j.exppara.2010.01.018. Epub 2010 Jan 28. PMID 20109451